CLINICAL TRIAL: NCT00370591
Title: Randomised, Double Blind, Parallel Group Study to Assess the Bronchodilative and Bronchoprotective Properties of SERETIDE DISKUS® Inhaler 50/100 mcg Twice Daily vs FLIXOTIDE® Inhaler 200 mcg Twice Daily
Brief Title: Study Of Airway Physiology In Adults. SERETIDE DISKUS® Inhaler and FLIXOTIDE® Inhaler Are Trademarks of GSK Croup of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM40104
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Inhaled corticosteroids; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Salmeterol/fluticasone propionate and fluticasone propionate

INTERVENTIONS:
Drug: Salmeterol/fluticasone propionate and fluticasone propionate

SUMMARY:
Comparison of two asthma treatments by lung function measures.

DETAILED DESCRIPTION:
Single centre, randomised, double-blind, comparator study to demonstrate superiority of salmeterol/fluticasone propionate combination product 50/100mcg bd over fluticasone propionate 100mcg bd with respect to improvements in airway physiology (sRAW) in adults with persistent asthma treated for 4 weeks.

ELIGIBILITY:
Inclusion:

* Physician documented diagnosis of asthma which has been present for at least 6 months.
* Receiving a total daily dose of 200-500mcg/day beclomethasone dipropionate or equivalent for at least 4 weeks prior to the start of the run-in period.

Exclusion:

* Has had 3 or more courses of oral corticosteroids in the 12 months previous to visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-12; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Specific airway resistance (sRAW kPa.L.s) measured before the study medication dose at the end of treatment (week 4)

SECONDARY OUTCOMES:
sRAW measured post-dose at Week 2 and week 4. % symptom-free days over Weeks 1-4. % symptom-free nights over Weeks 1-4. Type and frequency of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- [Derived] Houghton CM, Lawson N, Borrill ZL, Wixon CL, Yoxall S, Langley SJ, Woodcock A, Singh D. Comparison of the effects of salmeterol/fluticasone propionate with fluticasone propionate on airway physiology in adults with mild persistent asthma. Respir Res. 2007 Jul 14;8(1):52. doi: 10.1186/1465-9921-8-52. PMID 17629923
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAM40104 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register